CLINICAL TRIAL: NCT01845129
Title: Impact of Transcranial Direct Current Stimulation of the Motor Cortex on Language Functions in Residual Aphasia
Acronym: StimRAph
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Marcus Meinzer, Creutzfeldt Fellow, Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: RAPH_01EO0801
Record Dates: First submitted 2013-04-30; First posted 2013-05-03 (Estimated); Last update posted 2013-05-03 (Estimated); Status verified 2013-04

CONDITIONS: Residual Aphasia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- anodal tDCS (Experimental): atDCS will be administered for 20 minutes with 1 milliampere (1 mA) to the left primary hand motor cortex
  Interventions: Device: atDCS; Device: sham tDCS
- sham tDCS (Sham Comparator): sham tDCS will be administered to the left primary hand motor cortex
  Interventions: Device: atDCS; Device: sham tDCS

INTERVENTIONS:
Device: atDCS — atDCS will be delivered with a constant current of 1 mA during simultaneous resting-state (RS) and task-related (picture naming) functional magnetic resonance imaging (fMRI). The current will be turned on prior to the RS-fMRI scan and continues for 20 minutes.
Device: sham tDCS — During sham the current will be increeased and decreased in a ramp-like fashion (10 sec)

SUMMARY:
The present study assesses whether language functions in patients with residual post-stroke aphasia can be improved by transcranial direct current stimulation administered to the primary motor cortex in the language dominant (left) hemisphere.

DETAILED DESCRIPTION:
Patients will participate in two tDCS sessions (atDCS; sham) in a cross-over within subjects design. tDCS or placebo will be administered during simulatneous fMRI to assess neural signatures of the stimulation. Order of stimulation will be counterbalanced between subjects

ELIGIBILITY:
Inclusion Criteria:

* right handedness
* German native speaker
* cerebrovascular stroke in left hemisphere (>6 months)
* mild aphasia (according to Aachen Aphasia Test Battery Classification, Huber et al., 1983)
* residual anomia in naming test (>75 correct responses)

Exclusion Criteria:

* other current or previous neurological or psychiatric diseases
* alcohol or drug abuse
* MRI contraindication (e.g. magnetic metal, pacemaker, claustrophobia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2013-04; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
Response latency during picture naming task (max. 80) | Change in response latency between assessment 1 (week 1) and assessment 2 (week 2), assessments 1 and 2 are seperated by one week
  Subjects are assessed in a cross-over design. The primary outcome measure will be assessed twice in each subject, either during placebo ("sham) stimulation or active (anodal) stimulation with transcranial direct current stimulation. Order of stimulation will be counterbalanced across the group.

SECONDARY OUTCOMES:
Change in neural activity measured by functional magnetic resonance imaging | Change in fMRI activity between Assessment 1 (week 1) and Assessment 2 (week 2), assessments 1 and 2 are seperated by one week

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Meinzer, PhD, Principal Investigator — Charite, University Medicine, Neurology; Agnes Flöel, MD, Principal Investigator — Charite, University Medicine, Neurology
Locations (1):
- Charite, University Medicine, Dept. of Neurology, Berlin, State of Berlin, Germany